## DANIEL F. GOODMAN, MD GOODMAN EYE CENTER

## **Clinical Research Protocol**

# SAFETY AND EFFECTIVENESS OF THE PXL-PLATINUM 330 SYSTEM FOR CORNEAL CROSS-LINKING IN EYES WITH CORNEAL ECTASIA

| Protocol Number: | PXL-2211 |
|---|---|
| Version Date: | October 11, 2023 |
| Investigational Product: | Riboflavin 0.25% solution (Peschke-TE) |
| IND Number: | 146017 |
| Development Phase: | Phase 2 |
| Sponsor: | Name: Daniel F. Goodman, MD (Goodman Eye Center) Address: 2211 Bush Street, 2nd Floor, San Francisco, CA 95115 Telephone: 415-474-3333 Fax: 415-474-3939 Email: DGoodman@GoodmanEyeCenter.com |
| Principal Investigator: | Name: Daniel F. Goodman, MD (Goodman Eye Center) Address: 2211 Bush Street, 2nd Floor, San Francisco, CA 95115 Telephone: 415-474-3333 Fax: 415-474-3939 Email: DGoodman@GoodmanEyeCenter.com |
| Medical Monitor: | Name: Daniel F. Goodman, MD (Goodman Eye Center) Address: 2211 Bush Street, 2nd Floor, San Francisco, CA 95115 Telephone: 415-474-3333 Fax: 415-474-3939 Email: DGoodman@GoodmanEyeCenter.com |

| Approval: | |
|------------------------------------------|----------|
| PI or Sponsor Signature (Name and Title) | <br>Date |

## PROTOCOL AGREEMENT

I have read the protocol specified below. In my formal capacity as Principal Investigator, my duties include ensuring the safety of the study subjects enrolled under my supervision. It is understood that all information pertaining to the study will be held strictly confidential and that this confidentiality requirement applies to all study staff at this site. Furthermore, on behalf of the study staff and myself, I agree to maintain the procedures required to carry out the study in accordance with accepted GCP principles and to abide by the terms of this protocol.

| Protocol Number: | PXL-2211 | |
|---|---|---|
| Protocol Title: | Safety and Effectiveness of the PXL-Platinum 330 System for Cornea Cross-Linking in Eyes with Corneal Ectasia | |
| Protocol Date: | October 11, 2023 | |
| Investigator Signatu | re | <br>Date |
| Daniel F. Goodman,<br>Print Name and Title | , Principal Investigator | |

Site Name: Goodman Eye Center

Address: 2211 Bush Street, 2nd Floor

San Francisco, CA 95115

Telephone: 415-474-3333 Fax: 415-474-3939

## **TABLE OF CONTENTS**

| LI | ST OF ABBREVIATIONS | 5 |
|---|---|---|
| PF | ROTOCOL SYNOPSIS | 6 |
| 1. | BACKGROUND 1.1 Overview of Non-Clinical Studies 1.2 Overview of Clinical Studies 1.2.1 Conventional Crosslinking with Dresden Protocol 1.2.2 Accelerated or Pulsed Cross-Linking | 10<br>10<br>10<br>10<br>13 |
| 2. | RATIONALE 2.1 Risk/Benefit Assessment 2.2 Adverse Events | <b>15</b><br>15<br>17 |
| 3. | STUDY OBJECTIVES | 17 |
| 4. | STUDY DESIGN | 18 |
| 5. | STUDY OUTCOMES 5.1 Efficacy 5.2 Safety | <b>18</b><br>18<br>19 |
| 6. | STUDY POPULATION 6.1 Inclusion Criteria 6.2 Exclusion Criteria | <b>19</b><br>19<br>19 |
| 7. | <ul> <li>STUDY METHODS</li> <li>7.1 Subject Screening</li> <li>7.2 Subject Enrollment and Randomization</li> <li>7.3 CXL Treatment</li> <li>7.4 Retreatment Criteria</li> </ul> | 20<br>20<br>21<br>21<br>23 |
| 8. | INVESTIGATIONAL PRODUCT 8.1 Instructions for Use and Administration of Investigational Product (Riboflavin) 8.2 Formulation of Test Product 8.3 Supply of Study Drug at Site 8.4 Storage of Study Drug at Site 8.5 Study Drug Accountability 8.6 PXL Platinum 330 Illumination System | 23<br>24<br>24<br>24<br>24<br>24<br>25 |
| 9. | 9.1 VISIT 1- Screening Visit (Day -90 to Day 0) 9.1.1 Contact Lens Discontinuation 9.1.2 Keratoconus Severity 9.2 VISIT 2- Procedure Visit (Day 0) | 26<br>27<br>28<br>28<br>29 |

| | 9.3 VISIT 3- Day 1 Post-Op Visit (1-3 days Post-Op) | 29 |
|---|---|---|
| | 9.4 VISIT 4- Day 7/Week 1 Post-Op Visit (+/- 3 days) | 29 |
| | 9.5 VISIT 5- Month 1 Post-Op Visit (+/- 7 days) | 30 |
| | 9.6 VISIT 6- Month 3 Post-Op Visit (+/- 14 days) | 30 |
| | 9.7 VISIT 7- Month 6 Post-Op Visit (+/- 30 days) | 30 |
| | 9.8 VISIT 8- Month 12 Post-Op Visit/ End of Study Visit (+/- 30 days) | 31 |
| | 9.9 Early Withdrawal Visit | 31 |
| | 9.10 Early Withdrawal from Study | 32 |
| 10. | ADVERSE EVENT REPORTING | 32 |
| | 10.1 Adverse Event Definitions | 32 |
| | 10.2 Adverse Event Reporting and Documentation | 32 |
| | 10.2.1 Expected Non-Serious Ocular Adverse Events | 32 |
| | 10.3 Classification of Adverse Events by Severity | 32 |
| | 10.4 Classification of Adverse Event by Relationship | 33 |
| | 10.5 Serious Adverse Experiences (SAE) Definitions | 33 |
| | 10.6 Serious Adverse Event Reporting | 34 |
| 11. | PROTOCOL DEVIATIONS | 35 |
| 12. | DATA ANALYSIS AND STATISTICS | 36 |
| | 12.1 Sample Size | 36 |
| | 12.2 Accountability | 37 |
| | 12.3 Screening Data | 38 |
| | 12.4 Subject Characteristics | 38 |
| | 12.5.1 Visual Acuity | 38 |
| | 12.6 Secondary Efficacy Criteria | 38 |
| | 12.6.1 Keratometry | 38 |
| | 12.6.2 Manifest Refraction | 39 |
| | 12.6.3 Central Pachymetry | 39 |
| | 12.6.4 Endothelial Cell Count | 39 |
| | 12.6.5 Wavefront Aberrometry | 39 |
| | 12.7 Clinical Safety Endpoints | 40 |
| | 12.7.1 Adverse Events and Complications | 40 |
| | 12.7.2 Key Safety Parameters | 40 |
| | 12.8 Dropouts/Lost-to-Follow-Up | 40 |
| | 12.9 Interim Analysis | 40 |
| | 12.10 Sample Size and Randomization | 41 |
| 13. | DATA COLLECTION | 41 |
| | 13.1 Data Collection Instruments | 41 |
| 14. | ADMINISTRATIVE, ETHICAL, REGULATORY CONSIDERATIONS | 41 |
| | 14.1 Informed Consent | 41 |

| 14.2 Institutional Review Board | 41 |
|---------------------------------------------------------------|----|
| 14.3 Publications | 41 |
| 14.4 Investigator Responsibilities | 42 |
| 14.4.1 Medical and Safety Monitoring | 42 |
| APPENDIX A: Study Chart Flow | 43 |
| APPENDIX B: CFR 50.25 – Elements of Informed Consent | 46 |
| APPENDIX C: World Medical Association Declaration of Helsinki | 47 |
| APPENDIX D: References | 52 |

## LIST OF ABBREVIATIONS

**AE** adverse events

BCVA best corrected visual acuity
CDVA corrected distance visual acuity
CFR Code of Federal Regulations

CRF case report form
CXL corneal cross-linking
DMC data monitoring committee
DSMB data safety monitoring board
ECD endothelial cell density

**F** farenheit

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act of 1996

**ICF** informed consent form

ICH International Conference of Harmonisation

**IEC** Independent Ethics Committee

**IOP** intraocular pressure

IRB Institutional Review Board

**ITT** intent to treat

MRSE manifest refraction spherical equivalent

PI Principal Investigator

**PMD** pellucid marginal degeneration

**PP** per protocol

SAE serious adverse experience
SAP statistical analysis plan
UCVA uncorrected visual acuity

**UDVA** uncorrected distance visual acuity

**UVA** ultraviolet A

## **PROTOCOL SYNOPSIS**

| TITLE S | Cafety, and Effectiveness of the DVI Distingues 200 Contains for Orange - I |
|---|---|
| C | Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Cross-Linking in Eyes with Corneal Ectasia |
| SPONSOR D | Daniel F. Goodman, MD (Goodman Eye Center) |
| FUNDING ORGANIZATION | Daniel F. Goodman, MD (Goodman Eye Center) |
| NUMBER OF SITES | |
| | This study is being conducted to evaluate the safety and efficacy of the PXL-Platinum 330 system for performing corneal cross-linking. |
| de | Corneal collagen cross-linking is a modality that has been shown to elay or prevent corneal transplantation in patients with keratoconus nd/or post-refractive corneal ectasia. |
| ko<br>cı<br>si<br>si<br>aı<br>(s | n April 2016, the Avedro KXL system was approved by the FDA to treat eratoconus and post-refractive corneal ectasia via corneal ross-linking, using UVA light with riboflavin photosensitizer to trengthen corneal tissue. However, the Avedro KXL system can be a ignificant burden on patients, does not offer pulsed wave light delivery, nd was not approved for patients with other corneal thinning disorders such as pellucid marginal degeneration, immune-related corneal melts, on-progressive keratoconus). |
| p:<br>in | In contrast, the PXL-Platinum 330 system is less burdensome on patients, offers pulsed wave light delivery, and has shown effectiveness in treating other corneal thinning disorders not approved for indication with the Avedro KXL system. |
| STUDY DESIGN T | This is a randomized controlled trial with two parallel treatment arms. |
| (3 | reatment Group A: The cornea is irradiated with a pulsed UVA light 365 nm) at an irradiance of 4 mW/cm² between 10-15 seconds on and etween 10-15 seconds off for 45 minutes. |
| (3 | reatment Group B: The cornea is irradiated with a pulsed UVA light 365 nm) at an irradiance of 8 mW/cm² between 10-15 seconds on and etween 10-15 seconds off for 22.5 minutes. |
| <b>OBJECTIVE</b> po | o evaluate the safety and efficacy of the PXL Platinum 330 System for erforming corneal cross-linking (CXL) for the treatment of ectatic isorders. |
| SECONDARY To | o evaluate the safety and efficacy of the varying doses of power with |

| OBJECTIVE | pulsed (or fractionation) UV using the PXL Platinum 330 System. |
|---|---|
| NUMBER OF<br>SUBJECTS | 500 |
| SUBJECT<br>SELECTION<br>CRITERIA | Inclusion Criteria Subjects who have one or both eyes that meet criteria 1 and 1 or more of the following criteria (#'s 2-8) will be considered candidates for this study: |
| | 1. 10 years of age or older. |
| | Presence of central or inferior steepening. |
| | Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration. |
| | 4. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as: a. Fleischer ring b. Vogt's striae c. Decentered corneal apex d. Munson's sign e. Apical Corneal scarring consistent with Bowman's breaks f. Scissoring of the retinoscopic reflex Crab-claw appearance on topography |
| | 5. Steepest keratometry (Kmax) value ≥ 47.20 D. |
| | I-S keratometry difference > 1.5 D on the Pentacam map or topography map. |
| | 7. Posterior corneal elevation >16 microns. |
| | 8. Thinnest corneal point >300 microns. |
| | 9. Contact Lens Wearers Only: a. Removal of contact lenses for the required period of time prior to the screening refraction: Contact Lens Type Minimum Discontinuation Time Soft or Scleral 3 days Rigid gas permeable 2 weeks |

# **Exclusion Criteria** All subjects meeting any of the following criteria will be excluded from this study: 1. Eyes classified as either normal or atypical normal on the severity grading scheme. 2. Corneal pachymetry at the screening exam is <300 microns at the thinnest point in the eye(s) to be treated. 3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example: a. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthomeoeba, etc.) b. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure. 4. Pregnancy (including plan to become pregnant) or lactation during the course of the study. 5. A known sensitivity to study medications. 6. Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests. 7. Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing. TEST PRODUCT, The test product is Riboflavin (Peschke TE Riboflavin 0.25% ophthalmic DOSE, AND solution). The Riboflavin is administered in conjunction with a UVA light ROUTE OF via the PXL-Platinum 330 System. ADMINISTRATION **DURATION OF** The duration of subject participation is a total of 12 months for all study SUBJECT subjects following the CXL procedure visit. **PARTICIPATION** AND DURATION Duration of the study is ongoing until the 500 subject enrollment goal is OF STUDY met.

| CONCOMITANT<br>MEDICATIONS | There are no prohibited medications for enrolled subjects. |
|---|---|
| EFFICACY<br>EVALUATIONS | The primary efficacy endpoint will be Visual Acuity as defined by the absence of loss of UCVA and BCVA. |
| | The secondary efficacy endpoints will be changes from baseline for the following assessments: |
| | <ul> <li>Keratometry</li> <li>Manifest Refraction</li> <li>Central Pachymetry</li> <li>Endothelial Cell Count</li> <li>Wavefront Aberrometry</li> </ul> |
| SAFETY<br>EVALUATIONS | Primary safety evaluations will include a tabulation of unexpected and/or serious adverse events, patient symptoms, loss of visual acuity, slit lamp examination of the cornea and lens, and contact lens tolerance for contact lens wearers. |
| PLANNED<br>INTERIM<br>ANALYSIS | An interim analysis will be performed after all eyes complete the 3-month post-CXL procedure visit. |
| STATISTICS<br>Primary Analysis<br>Plan | The primary analysis plan will include a two sample t-test, a repeated measure analysis of variance, and descriptive statistics. |
| Rationale for<br>Number of<br>Subjects | Enrolling 202 eyes in each treatment group will enable the detection of a 20% difference in UCVA for both genders. The sample size is adjusted for a 10% rate of discontinued and lost-to-follow-up eyes. |

## 1.BACKGROUND

This study is being conducted to evaluate the safety and effectiveness of the PXL Platinum 330 system for performing corneal cross-linking (CXL) for the treatment of ectatic disorders. The PXL Platinum 330 system is a combination product consisting of a UVA 365 nm wavelength light source (PXL Platinum 330 Illumination System) and riboflavin (Peschke TE Riboflavin 0.25% ophthalmic solution). The riboflavin is administered in conjunction with the UVA light and acts as a photosensitizer.

The PXL Platinum 330 treatment is intended to induce corneal cross-linking to improve the biomechanical properties of the cornea by strengthening the corneal tissue in the anterior stroma. Corneal cross-linking is performed by pretreating the cornea with riboflavin 0.25% ophthalmic solution beginning 30 minutes before UVA light exposure to saturate the corneal tissue with the riboflavin photosensitizer. The cornea is then irradiated with a pulsed UVA light (365 nm) at an irradiance of either 4 mW/cm² between 10-15 seconds on and between 10-15 seconds off for 45 minutes or 8 mW/cm² between 10-15 seconds on and between 10-15 seconds off for 22.5 minutes – both producing a maximum energy dose of 5.4 J/cm². Exposure of the cornea to this combination of UVA light (365 nm; 5.4 J/cm² energy dose) after topical administration of riboflavin 0.25% has been shown to induce cross-linking of the corneal collagen fibrils with a resultant increase in tensile strength and diameter of the collagen fibrils. Clinically, cross-linking has been shown to stabilize the corneal curvature in eyes with progressive keratoconus with no significant change in the refractive index of the cornea. It is unknown however if varying doses of power with pulsed (or fractionation) UV offers greater efficacy and safety.

## 1.1 Overview of Non-Clinical Studies

Preclinical investigations have been performed to: (1) determine the optimal photosensitizing agent/dosage and irradiance/exposure time for cross-linking; (2) characterize the biomechanical and biochemical effects of cross-linking on corneal collagen tissue using rabbit, porcine, and human corneal tissue models; and, (3) determine toxicity to keratocytes and endothelial cells.

#### 1.2 Overview of Clinical Studies

## 1.2.1 Conventional Crosslinking with Dresden Protocol

UVA/riboflavin corneal collagen cross-linking was first used clinically in 1998. (Unless specified otherwise, the treatments referenced below in this subsection all used UVA light (365 nm, 3 mW/cm² at 30 minutes) with photosensitizing riboflavin 0.25% (10 mg in 10 mL Dextran-T-500 20% solution applied after a central corneal abrasion, beginning at least 5 minutes before irradiation and continuing every 5 minutes during irradiation.)

Wollensak et al. treated 23 eyes of 22 patients to evaluate the effect of cross-linking on patients with moderate or advanced keratoconus. The mean preoperative maximum K-value (Kmax) was 50.93 D, and the mean preoperative progression of Kmax was 1.42 D

(±1.18 D) in the 6 months before cross-linking. After cross-linking, there was a mean decrease in Kmax of 2.01 D (p=0.001) with follow-up of 3 to 47 months (mean 23.2 ±12.9 months). In five of the untreated contralateral eye controls, the mean Kmax progressed an average of 1.48 D in the first year after cross-linking was performed in the contralateral eyes. Best spectacle corrected visual acuity (BSCVA) improved by an average of 1.26 lines (p=0.026) and manifest refraction spherical equivalent (MRSE) improved by an average of 1.14 D (p=0.03) in the treated eyes. No adverse events occurred. The postoperative healing process was unremarkable except for slight transient stromal edema during the first 3 postoperative days. Corneal and lens transparency, intraocular pressure (IOP), and endothelial cell density (p=0.45) were unchanged after treatment compared to baseline.

Similarly, Caporossi et al. reported a 3.6 line increase in uncorrected visual acuity (UCVA), a 1.66 line improvement in BSCVA, a mean reduction in Kmax of 2.1 D (±0.13), and a 2.5 D reduction in MRSE at 3 months after cross-linking in a series of 10 eyes in 10 patients with progressive keratoconus. There were no changes in endothelial cell density or IOP.<sup>2</sup>

Patients treated in an ongoing clinical study at the University of Dresden (Dresden, Germany), have experienced outcomes similar to those reported by Wollensak.<sup>3</sup> A preliminary analysis of the Dresden keratometry data shows a 1.25 D reduction in maximum corneal curvature (K<sub>max</sub>) in those eyes that have reached the 6-month evaluation time point. Progressively increasing corneal curvature is a hallmark of keratoconus and corneal ectasia. Based on the preliminary analysis of the Dresden data, corneal curvature progression is halted in this series of patients. The effect is significant 5 years after the CXL treatment and the trend continues to be observed as long as 7 years after cross-linking.

Table 1: Change in Maximum Corneal Curvature (Kmax) in Eyes treated with CXL

| Time | N | Baseline<br>Mean<br>Kmax<br>(diopters) | Post-CXL<br>Mean Kmax<br>(diopters) | Difference<br>in Kmax<br>(diopters) | Kmax<br>Percent<br>Difference<br>(%) | Kmax<br>Difference<br>(p<0.05) | Kmax %<br>Difference<br>(p<0.05) |
|---|---|---|---|---|---|---|---|
| Baseline | 365 | 53.6044 | | | | | |
| 6 Months | 196 | 53.9003 | 52.6523 | -1.24801 | -1.83121 | 0.001013 | 0.002256 |
| 1 Year | 136 | 53.7790 | 52.3346 | -1.44449 | -2.35446 | 0.000025 | 0.000039 |
| 2 Years | 60 | 54.0197 | 52.4340 | -1.58567 | -2.52731 | 0.001214 | 0.001250 |
| 4 Years | 30 | 53.4627 | 50.7030 | -2.75967 | -4.58245 | 0.000396 | 0.000342 |
| 5 Years | 13 | 52.2777 | 50.0723 | -2.20538 | -3.78418 | 0.020667 | 0.019656 |
| 6 Years | 5 | 50.6400 | 48.1740 | -2.46600 | -4.81223 | 0.064549 | 0.067719 |
| 7 Years | 4 | 52.3825 | 49.4500 | -2.93250 | 05.48322 | 0.057697 | 0.056259 |
| 8 Years | 1 | 47.3400 | 47.1400 | -0.20000 | -0.42248 | | |

Kohlhaas presented results for 127 of these eyes at the 2005 Congress of the German-Language Society for Intrakularlinsen Implantation and Refraktive Surgery with a follow-up of up to 60 months. Progression of keratoconus was stopped in all the eyes, and 81.7% of them showed a mean decrease of 2.87 D in Kmax. No opacification of the lens or change in endothelial cell density was seen in any patient.

Long term follow-up results in a subset of 60 eyes in the Dresden Clinical Study that underwent cross-linking 3-5 years prior confirm the lasting effects of cross-linking in that there has been no progression of keratoconus in any of the eyes and 51.2% (31/60) of the eyes have a slight reversal and flattening of the Kmax.<sup>4</sup> Kohlhaas, et al. also reported a patient who developed bilateral keratectasia at 4 weeks after LASIK and underwent UVA/riboflavin cross-linking 6 months later.<sup>5</sup> In this case, corneal topography remained stable for 18 months after cross-linking.

Fifty eyes in 36 patients have been enrolled in an Australian randomized study of observation-only control versus cross-linking in eyes with progressive keratoconus. Maximum K-readings taken before and at 3 and 6 months after cross-linking showed a mean decrease of -1.10 diopters and -1.39 diopters in the treatment group. In contrast, the untreated control eyes show a statistically significant 0.70 D and 0.78 D increase in K-readings at 3 and 6 months after randomization. The treatment group also showed a mean 2.2-line improvement in BSCVA at 3 and 6 months, while BSCVA in the control group worsened. Similar to the Dresden experience, these data lead to the conclusion that corneal cross-linking halts, and may even reverse, the progression of keratoconus.

**More recent studies** confirm long-term improvement in eyes treated with cross-linking, including a 10 year follow-up study as well as a crossover study, and 3 trials in pediatric populations. <sup>7,8,9,10,11,12,13,14,15,16,17</sup>

With respect to the use of the Dresden protocol with the Peschke system, the relevant papers include:

- Corneal Cross-Linking and Safety Issues
   Open Ophthalmo/ J. 2011; 5: 14-16. Eberhard S et al.

   The authors analyzed the current treatment protocol regarding safety during CXL with the riboflavin/UVA (370 nm) approach. When the corneal stroma thickness is at least 400 microns, a homogenous irradiance of UV light of 3mW/cm² for 30 min at 370 nm with the application of 0.1% riboflavin didn't damage either corneal endothelium or deeper structures such as lens and retina.
- Prospective, randomized, double-blind trial to investigate the efficacy and safety of corneal cross-linking to halt the progression of keratoconus. BMC Ophthalmology 2015; 15:78. Stefan Lang et al.

The efficacy and safety of corneal cross-linking were investigated in a randomized, blinded, placebo controlled, multicenter trial. Fifteen eyes were randomized to the treatment group (corneal epithelial removal, 0.1% riboflavin, UVA 370 nm at 3mW/cm² for 30 min) and 14 to the control group (no epithelial removal, fluorescein drops, visible blue light for 30 min). Follow-up averaged 1098 days. The treatment group showed a decrease in corneal refractive power (on average 0.35 diopters/year) while the controls showed an increase of 0.11 diopters/year. However, some of the treated patients still progressed, whereas some controls improved. The change in visual acuity did not show a statistically significant difference between the two groups.

## 1.2.2 Accelerated or Pulsed Cross-Linking

Pulsed cross-linking seems to be able to enhance functional and structural outcomes due to improved oxygen bioavailability during the crosslinking reaction. The stromal demarcation line (commonly accepted as a marker of depth of biomechanical strengthening) was deeper with pulsed cross-linking in 2 studies (Moamarco et al. LRS 2015 and Mazzotta et al. Eye 2014). Mazzotta et al.'s 1 year results (J. Ophthalmol 2014) show that pulsed crosslinking achieved a 1.2 diopter reduction in corneal keratometry, whereas continuous light cross-linking only resulted in 0.13 diopter reduction.

With respect to the use of accelerated or pulsed crosslinking using the Peschke system, the relevant studies include:

# • Accelerated (18mW/cm²) Corneal Collagen Cross-Linking for Progressive Keratoconus.

Cornea. 2015 Nov;34(11):1427-31. Alnawaiseh M et al.

The charts and anterior segment data of 20 patients (28 eyes) who were treated with accelerated corneal collagen cross-linking (18 mW/cm²; 5 minutes) were reviewed. The mean follow-up time was 21.7 months. It found a significant reduction (improvement) of Kmax (the steepest radius of curvature of the anterior corneal surface) and stabilization of corrected distance visual acuity (CDVA) with no reported complications.

## Accelerated (9-mW/cm²) corneal collagen crosslinking for keratoconus- A 1-year follow-up.

Cornea. 2014 Aug;33(8):769-73. Elbaz U et al.

Sixteen mild-moderate keratoconus-affected eyes (14 patients) underwent an accelerated crosslinking (irradiance of 9 mW/cm²; 10 minutes). At either 6 or 12-month follow-up, no statistically significant changes were found in the mean CDVA, mean refractive cylinder, or mean manifest refraction spherical equivalent. There was an improvement in the uncorrected distance visual acuity (UDVA); a gain of 0.13 logarithm of the minimum angle of resolution lines in the mean UDVA (P = 0.012). Ksteep, Kflat, average K (Km), corneal astigmatism (Kcyl), and maximal curvature reading at the corneal apex (Kmax) were stable.

• Safety of high-intensity corneal collagen crosslinking

J Cataract Refract Surg. 2014 Aug;40(8):1337-40. George Kymionis et al.

Ten eyes (9 patients) underwent corneal cross-linking with 9mW/cm² irradiance for 10 minutes. Three months after procedure, endothelial cell density (ECD) did not change and CDVA improved but the improvement wasn't statistically significant. No eye lost lines of CDVA. The mean steep K readings decreased significantly.

One-year outcomes of conventional and accelerated collagen crosslinking in progressive keratoconus
 SciRep. 2015 Sep 25;5:14425. Vanissa Chow et al.
 Nineteen eyes in each group underwent conventional (3 mW/cm², 365-nm UVA, 30 minutes) or accelerated (18 mW/cm², 365-nm UVA, 5 minutes) collagen crosslinking. One year postoperatively, there were no inter-group differences in keratometry, UCVA, and best corrected visual acuity (BCVA).

- Evaluation of Corneal Stromal Demarcation Line Depth Following Standard and a Modified-Accelerated Collagen Cross-linking Protocol
   Am J Ophthalmol. 2014 Oct;158(4):671-675. George Kymionis et al.
   Twenty-six eyes were treated for 30 minutes with 3 mW/cm² UVA, while 26 eyes were treated for 14 minutes with 9 mW/cm² UVA. One month postoperatively, corneal stromal demarcation line depth was assessed using AS-OCT with no significant difference between the two groups.
- Safety profile of accelerated corneal cross-linking versus conventional cross-linking: a comparative study on ex vivo-cultured limbal epithelial cells BrJ Ophthalmol. 2015 Feb;99(2):272-80.Rohit Shetty et al.
  Day 14 cultured limbal epithelial cells (LECs) were either unexposed (control) or exposed to different intensities of UVA irradiance for different durations (3 mW for 30 min, 9 mW for 10 min, 18 mW for 5 min and 30 mW for 3 min) in the presence and absence of riboflavin. When the apoptotic status was evaluated through quantitative real-time PCR, vital staining, immunofluorescence staining and fluorescence-activated cell sorting, it was shown that the 30 mW UVA irradiation used in accelerated corneal cross-linking appears to be safe on cultured LECs in comparison with 3 mW used in corneal cross-linking.
- Corneal stroma demarcation line after standard and high-intensity collagen crosslinking determined with anterior segment optical coherence tomography J Cataract Refract Surg. 2014 May;40(5):736-40. George Kymionis et al. Nine eyes were treated for 30 minutes with 3 mW/cm² UVA and 12 eyes were treated for 10 minutes with 9 mW/cm² of UVA. One month after procedure, the corneal stroma demarcation line was significantly deeper after a 30-minute 3 mW/cm² UVA treatment than after a 10-minute 9 mW/cm² of UVA irradiation.

# 2. RATIONALE

Keratoconus is a naturally occurring ocular condition characterized by progressive thinning and steepening of the central cornea, resulting in increasing myopia, irregular astigmatism, and eventual loss of best spectacle-corrected visual acuity. Rigid contact lenses can be used to improve visual acuity in many patients, but keratoconus frequently progresses to the point that corneal transplantation is required to restore useful vision. Keratoconus may recur following corneal transplantation and require further transplant surgery.

Together, keratoconus and post-refractive corneal ectasia are the second most frequent indication for corneal transplantation, accounting for about 15% of the corneal transplants performed in the United States. Corneal transplantation has inherent risks that could result in permanent loss of vision and significantly impact the patient's quality of life during the surgical recovery phase, with lost work time and often permanent changes in lifestyle. Any modality, such as corneal collagen cross-linking, that can delay or prevent corneal transplantation in patients with these conditions is of great benefit.

Corneal collagen cross-linking using UVA light with riboflavin photosensitizer to strengthen corneal tissue was approved by the FDA in April 2016 with the Avedro KXL system for slowing or stopping the progression of keratoconus and post-refractive surgery ectasia. However, patients with other corneal thinning disorders (pellucid marginal degeneration, immune-related corneal melts, non-progressive keratoconus) were not included in the approved indication. Further, the Avedro KXL system is a significant burden on patients and clinics due to requirement for epithelial scraping (which increases pain, infection risk, and scarring risk), time necessary to perform the procedure, expense, and lack of reimbursement. Lastly, the approved system does not offer pulsed wave light delivery, which seems to improve outcomes after crosslinking in keratoconus due to improved oxygen availability.<sup>21,22,23</sup>

Clinical applications of corneal cross-linking include treatment or prophylaxis of conditions distinguished by corneal thinning, such as post-LASIK ectasia, keratoconus, and pellucid marginal degeneration.

## 2.1 Risk/Benefit Assessment

Riboflavin, also known as Vitamin B2, is a naturally occurring photosensitizer. It is the precursor of flavin mononucleotide (FMN) and flavin adenine dinucleotide (FAD), two coenzymes that are crucial for the metabolism of carbohydrates, fats and proteins into energy. Riboflavin is an essential constituent of all living cells. It is water soluble and only a trace amount is found in the human body. Riboflavin is water-soluble and is non-toxic; it is used as a coloring agent in food and pharmaceuticals. The intake of riboflavin from food and diet supplements ranges from 4 to 10 mg a day. No adverse effects have been associated with high intakes of riboflavin from food or supplements.

Pharmacokinetic studies have shown that the maximal amount of riboflavin that is absorbed after a single oral dose is 27 mg, regardless of the amount in excess of this that is ingested. Excess riboflavin is excreted in urine and, since it is not a fat-soluble vitamin, is not stored in fat or other body tissues. No upper limit for riboflavin uptake has been established by the Food and Nutrition Board of the Institute of Medicine of the National Academy of Sciences due to insufficient human and animal data. A risk assessment performed by the UK government has determined that a total intake of 43 mg is not expected to result in any adverse effects.<sup>24</sup>

The standard concentration of riboflavin used in the riboflavin/UVA treatment is 0.1%. The maximum amount of riboflavin to which a patient is exposed during treatment is estimated to be 1.6 mg based on the volume of one drop being 0.05 ml and 1 drop being instilled every 2 minutes for 30 minutes before, and 30 minutes during, UVA light irradiation (32 drops). This is below the 43 mg "safe" limit by an order of magnitude.

The potential cytotoxicity of UVA light and the UVA/riboflavin exposure on keratocytes and endothelial cell function have been characterized in a series of in vitro experiments. In each of these experiments, UVA exposure (370 nm, 30 minutes) and riboflavin (0.025% solution; equivalent to the corneal concentration after diffusion of a 0.1% solution) were administered to mimic conditions of clinical usage. Irradiance levels were varied to determine the irradiance threshold for cytotoxic effects. Keratocyte toxicity was evaluated in porcine keratocyte cell cultures after exposure to riboflavin alone, UVA light alone (irradiance range 2 to 9 mW/cm<sup>2</sup>) and UVA light plus riboflavin (irradiance range 0.4 to 1 mW/cm<sup>2</sup>)<sup>25</sup>. Riboflavin alone had no cytotoxic effect on keratocytes. The cytotoxic threshold for inducing cellular necrosis or apoptosis was 5 mW/cm<sup>2</sup> for UVA light alone and 0.5 mW/cm<sup>2</sup> for the UVA/riboflavin treatment. Using the Lambert-Beer equation, in human corneas the cytotoxic keratocyte UVA irradiance of 0.5 mW/cm<sup>2</sup> is reached at a stromal depth of 300 microns. The potential for endothelial cell toxicity was evaluated on endothelial cell cultures obtained from porcine cornea that were exposed to riboflavin alone and to various UVA irradiances (range 0.1 to 1.6 mw/cm<sup>2</sup>) with and without riboflavin.<sup>26</sup> An abrupt cytotoxic threshold was observed at an irradiance of 4 mW/cm<sup>2</sup> for UVA light alone and was tenfold lower with an irradiance threshold of 0.35 mW/cm<sup>2</sup> for the UVA/riboflavin treatment.

No endothelial cell damage was observed in the cells treated with riboflavin alone. Endothelial cell damage is believed to be due to oxidative damage caused by the oxygen reactive free radicals (singlet oxygen, superoxide anion, hydrogen peroxide) that are generated by the UV light.<sup>27</sup>

The lower cytotoxic thresholds observed for the UVA/riboflavin combination in the keratocyte and endothelial cell toxicity studies is consistent with the increase in UVA absorption in the anterior cornea in the presence of riboflavin. For example, 94% of incident UVA light is absorbed in the anterior 400 microns of the corneal stroma in the presence of riboflavin, as depicted in the graph below, whereas only 32% is absorbed within that depth in the absence of riboflavin.<sup>28</sup>

#### 2.2 Adverse Events

Adverse events have been reported after cross-linking. Corneal edema occurred in an eye with a pretreatment corneal thickness of <400 microns, presumably caused by UV damage to the corneal endothelium.<sup>29</sup> Using confocal microscopy, Mazotta et al. evaluated 10 patients treated with UVA/riboflavin for progressive keratoconus and found normal epithelial morphology and an absence of subepithelial stromal nerve fibers in the central irradiated area at 5 days after cross-linking.<sup>30</sup> Nerve regeneration was observed at 1 month and nerve fiber recolonization was complete at 6 months with restoration of corneal sensitivity. No changes were observed in the peripheral untreated area at any time. Recently, Seiler et al. described a thin corneal stromal demarcation line that was detectable by slit lamp microscopy at a depth of -300 microns 2 weeks after cross-linking in 14 of 16 eyes evaluated.31 This demarcation line is believed to be due to a difference in the refractive index or reflection properties of untreated and cross-linked corneal stroma. When epithelial thickness (~50 microns) is taken into account, the 300 micron demarcation line observed by Seiler et al. is consistent with the studies and theoretical principles that the selected parameters for UVA/riboflavin treatment produce maximal cross-linking to a depth of about 200 microns and that 94% of the UVA light is absorbed in the anterior 300 microns of corneal stroma without injury to the endothelium. Hafezi et al. recently published the results of corneal collagen cross-linking in 10 eyes of 10 patients who had ectasia after prior LASIK surgery.<sup>32</sup> Anterior stromal haze was observed in the early postoperative period in all 10 eyes, with the corneas completely clear at the 12-month evaluation. This anterior stromal haze is similar to the subepithelial haze that is seen with photorefractive keratectomy (PRK) procedures, but the haze after cross-linking is not subepithelial in nature. The anterior stromal haze has also been reported anecdotally by the Australian investigators as a typical occurrence after cross-linking that disappears within 3 to 6 months after the procedure and is thought to be related to keratocyte apoptosis and regeneration after cross-linking.33

Rare cases of persistent epithelial defect or corneal infection have been reported after crosslinking, typically after epithelium-off crosslinking which entails scraping of epithelium, allowing access for bacteria or other microorganisms to invade the corneal stroma.

Additionally, common non-serious adverse events expected to be observed in the eye or eye(s) within the first few days and up to four weeks after the procedure include the following: pain, photophobia, foreign body sensation, dryness, irritation, and blurred vision.

#### 3. STUDY OBJECTIVES

The primary objective of this study is to evaluate the safety and efficacy of corneal collagen cross-linking (performed using the PXL-Platinum 330 system) for treating corneal curvature and biomechanical anomalies associated with corneal ectatic conditions (e.g., progressive or non-progressive keratoconus, pellucid marginal degeneration, and post-LASIK corneal ectasia).

Secondary study objectives include an evaluation of the safety and efficacy of varying doses of power with pulsed (or fractionation) UV using the PXL Platinum 330 System.

#### 4. STUDY DESIGN

This is a prospective, double-armed, randomized, single-site study to determine the safety and effectiveness of the PXL Platinum 330 system for performing corneal collagen cross-linking (CXL) in eyes with corneal ectasia. Subjects with a history of keratoconus, forme-fruste keratoconus, pellucid marginal degeneration, post-LASIK ectasia, diurnal fluctuation post-radial keratotomy, and Terrien's marginal degeneration will be evaluated initially for suitability as a candidate for CXL.

Subjects that are candidates for CXL will be asked to participate in this study and will undergo the required screening procedures to determine study eligibility. Informed consent will be obtained from each subject before performance of any required study procedures that are not part of the Investigator's routine examination. After completing the screening procedures, screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and no exclusion criteria will be entered into the study.

Subjects will be randomized into one of two treatment groups:

- <u>Treatment Group A:</u> 4 mW/cm<sup>2</sup> between 10-15 seconds on and between 10-15 seconds off for 45 minutes
- <u>Treatment Group B:</u> 8 mW/cm<sup>2</sup> between 10-15 seconds on and between 10-15 seconds off for 22.5 minutes

Total duration of subject participation will be twelve months after the CXL procedure visit. The duration of the study will be extended for those subjects who have received retreatment or for subjects who elect to have CXL treatment in an untreated fellow eye.

Total duration of the study is expected to be ongoing until the 500 subject enrollment goal is met.

#### 5. STUDY OUTCOMES

## 5.1 Efficacy

The primary efficacy endpoint is visual acuity, both UCVA and BCVA. Study success is defined by the absence of loss of UCVA and BCVA. Secondary efficacy endpoints include the evaluation of additional measurements of corneal curvature, as measured by maximum keratotomy ( $K_{max}$ ) and mean keratotomy ( $K_{mean}$ ) in the randomized eye(s). Study success is defined as the absence of corneal steepening defined as an increase of  $K_{max}$  or  $K_{mean}$  of  $\geq 0.5$  diopters from Day 0 to 12 months in the treated eye(s). Secondary efficacy measurements will also include: pachymetry, diopters of astigmatism as measured by keratometric cylinder,

posterior corneal elevation, manifest refraction, endothelial cell count, and wavefront aberrometry.

## 5.2 Safety

Safety assessments will include a tabulation of unexpected and/or serious adverse events, patient symptoms, loss of visual acuity, slit lamp examination of the cornea and lens, and contact lens tolerance for contact lens wearers.

## 6. STUDY POPULATION

This study is a single-center study that will be conducted over 5 years. Up to 500 subjects with corneal ectatic conditions who meet the inclusion and exclusion criteria will be eligible for participation in the study.

#### 6.1 Inclusion Criteria

Subjects who have one or both eyes that meet criteria 1 and 1 or more of the following criteria (#'s 2-8) will be considered candidates for this study:

- 1. 10 years of age or older
- 2. Presence of central or inferior steepening
- 3. Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
- 4. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as:
  - a. Fleischer ring
  - b. Vogt's striae
  - c. Decentered corneal apex
  - d. Munson's sign
  - e. Apical Corneal scarring consistent with Bowman's breaks
  - f. Scissoring of the retinoscopic reflex Crab-claw appearance on topography
- 5. Steepest keratometry (Kmax) value ≥ 47.20 D
- 6. I-S keratometry difference > 1.5 D on the Pentacam map or topography map
- 7. Posterior corneal elevation >16 microns
- 8. Thinnest corneal point >300 microns
- 9. Contact Lens Wearers Only:
  - a. Removal of contact lenses for the required period of time prior to the screening refraction:

**Contact Lens Type Minimum Discontinuation Time**Soft or Scleral 3 days

Rigid gas permeable 2 weeks

#### 6.2 Exclusion Criteria

All subjects meeting any of the following criteria will be excluded from this study:

- 1. Eyes classified as either normal or atypical normal on the severity grading scheme.
- 2. Corneal pachymetry at the screening exam is <300 microns at the thinnest point in the eye(s) to be treated.
- 3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:
  - a. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthomeoeba, etc.)
  - b. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
- 4. Pregnancy (including plan to become pregnant) or lactation during the course of the study
- 5. A known sensitivity to study medications
- 6. Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
- 7. Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing.

#### 7. STUDY METHODS

#### 7.1 Subject Screening

Subjects will be screened by the Investigator or his/her designee based upon the following criteria that are detailed in the case report forms to be utilized for the screening visit:

- Demographics
- Contact Lenses History
- Medical History
- Ocular History
- Medication History (Concomitant Medications)
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry
- Pentacam
- Corneal Topography by TMS-4
- IOP
- Endothelial Cell Count
- OCT K
- Wavefront Aberrometry
- Belin ABCD Progression

- Slit Lamp Examination
- Dilated Fundus Exam (if not done in the past 12 months)
- Inclusion/Exclusion Criteria

Once all of the study requirements for enrollment have been reviewed and determination that the eligibility criteria have been met, the Investigator will enroll the subject into the study.

## 7.2 Subject Enrollment and Randomization

Upon enrollment in the study, the study subject will be randomly assigned to one of the two treatment groups in a 1:1 ratio using the randomization app titled "Random".

On the day of the CXL procedure, an interim medical history, ocular history, and medication history will be obtained to determine whether any events or changes in health status have occurred that would preclude the subject from undergoing CXL treatment at the scheduled time or from participating in the study. Measurements from the complete eye examination that were performed during screening and/or routine examination may be repeated, at the discretion of the investigator, to provide accurate baseline measurements.

If the results of any repeat measurements performed on the CXL treatment day fail to meet eligibility criteria, the CXL treatment will be postponed or the subject will be dropped from the study.

Prior to the CXL treatment, the staff will confirm that the informed consent form for the study has been signed.

#### 7.3 CXL Treatment

Enrolled subjects will be prepared for CXL treatment in accordance with the instructions for use in the PXL Platinum 330 Illumination System Operator's Manual.

## Surgical Procedure for CXL

CXL will be performed on an outpatient basis using the PXL Platinum 330 System (UVA light source and riboflavin solution). All use of the PXL Platinum 330 System will be in accordance with the protocol and the general instructions provided by the manufacturer in the PXL Platinum 330 Operator's Manual.

A summary of the general technique for performing CXL is summarized below. CXL procedures used for each subject will be documented on the source documents. Selected treatment information, including the riboflavin administration, irradiance settings, and duration of irradiation exposure will be documented.

## **Subject Preparation and Riboflavin Administration**

Eyes undergoing CXL will have topical anesthetic administered. After topical anesthesia, the surgeon or trained designee will apply topical riboflavin onto the cornea (1 drop every 1 minute for approximately 30 minutes with trans-epithelial treatment).

The duration of riboflavin application will vary and will be determined by the physician's determination by biomicroscopic (slit lamp) exam that complete corneal stromal saturation is achieved - which varies from patient to patient. Methylcellulose sponges and "corneal light shields" will be used to enhance permeability.

If the corneal stroma is not saturated adequately, riboflavin will continue to be instilled 1 drop every 1 minute for an additional 10 minutes, and the stroma will be rechecked for saturation. This process will be repeated as necessary.

#### **CXL Procedure**

After the riboflavin pre-treatment regimen is complete and corneal stromal saturation is confirmed, the eye will be aligned under the PXL Platinum 330 light (the treatment plane will be at the correct working distance from the PXL Platinum 330 beam aperture when the border of the projected beam is in sharp focus – 50 mm). The correct aperture setting will be 12 mm and the eye will be irradiated at either 4 mW/cm², with pulsed mode (between 10-15 seconds on, 10-15 seconds off) for 45 minutes (Treatment Group A) or 8 mW/cm² with pulsed mode (between 10-15 seconds on, 10-15 seconds off) for 22.5 minutes (Treatment Group B). In both groups, the total energy dose will be 5.4 J/cm². At the end of the treatment, the UV light source will automatically switch to the off position. The operator will keep track of irradiation time independently to confirm the actual treatment time.

Topical anesthetics will be administered as needed to maintain patient comfort during the CXL procedure.

The eye will be examined at a slit lamp; a drop of antibiotic will be placed. A bandage contact lens will be placed, to be worn until seen by the physician the next morning.

#### **UVA Light**

Prior to the first treatment of the day, the PXL Platinum 330 illumination system will be assembled and tested according to the manufacturer's instructions. The UV irradiance dose is the product of the irradiance intensity and the exposure time. The intensity is a fixed parameter of the device. It is checked during the light test and cannot be changed by the user.

## **Postoperative Care**

Prescriptions for postoperative medications and written postoperative instructions will be given to each subject and reviewed prior to discharge. The following postoperative eye drops will be prescribed:

- 1. Topical antibiotic x 7 days
- 2. Topical steroid drop x 7 days
- 3. Preservative-free artificial tears hourly while awake for at least 48 hours

All postoperative eye drop usage will be recorded in the subject's chart. Other prescription or nonprescription medications, including pain medication, may be taken as needed throughout the study.

Subjects will remain in the clinic until the CXL treatment has been completed and the investigator determines that it is safe for the subject to be discharged from the clinic. Generally, the average time from arrival to discharge is approximately 2 hours.

#### 7.4 Retreatment Criteria

The CXL treatment is intended to be a one-time treatment. If progression of  $K_{max}$  or  $K_{mean}$  defined as an increase of 1.0 diopters or more is observed at 6 or 12 months, the subject will be offered retreatment.

If a subject receives crosslinking retreatment with the study device, the duration of the study will be extended for 6 months after the retreatment. The subject will receive additional study visits according to the following schedule:

- Retreatment Operative (Day 0)
- Retreatment Day 1 (1 to 3 days post procedure)
- Retreatment Week 1 (+/- 3 days)
- Retreatment Month 1 (3 to 5 weeks)
- Retreatment Month 3 (10 to 14 weeks)
- Retreatment Month 6 (21 to 30 weeks)
- Retreatment Month 12 (47 to 55 weeks)

The procedures and assessments at the retreatment visits are the same as those which take place at the original post-op visits at the same time points. If a patient is retreated and the timing of the visit windows allows, the retreatment visits may be combined with the post-op visits from the original cross-linking procedure (e.g. if a patient is retreated shortly after their 6 month post-op, their 6 month retreatment post-op can be combined with their 12 month post-op from the original procedure).

## **Post-Study Procedures**

Subjects will be discharged from the study after the 12-month follow-up examination is complete. Clinically significant abnormalities will be followed until the abnormality returns to acceptable limits or there is an adequate explanation for the abnormality.

## **Blinding**

Due to the objectives of the study, the PI will not perform any postoperative exams to ensure blindness of the study. The study blind will be broken on completion of the clinical study and after the study database has been locked. During the study, the blind may be broken only in emergencies when knowledge of the patient's treatment group is necessary for further patient management.

#### 8. INVESTIGATIONAL PRODUCT

The test product is Riboflavin (Peschke TE Riboflavin 0.25% ophthalmic solution).

The Riboflavin solution is obtained from: Peschke-MediTrade GmbH Chaesigass 6a 6331 Huenenberg, Switzerland

The Riboflavin is administered in conjunction with a UVA light via the PXL-Platinum 330 System.

## 8.1 Instructions for Use and Administration of Investigational Product (Riboflavin)

Riboflavin will be administered according to the instructions provided by the manufacturer. One drop of Riboflavin 0.25% ophthalmic solution will be instilled topically in the eye every 1 minute for 15-30 minutes, until the physician determines by slit lamp biomicroscopy that the corneal stroma has been saturated, which varies from patient to patient (riboflavin emits a brilliant auto-fluorescence easily detectable in the cornea stroma). Methylcellulose sponges and "corneal light shields" will be used to enhance permeability. If the corneal stroma is not saturated adequately, riboflavin will continue to be instilled 1 drop every 1 minute for an additional 10 minutes, and the stroma will be rechecked for saturation. This process will be repeated as necessary.

#### 8.2 Formulation of Test Product

The riboflavin solution is an isotonic (0.9%) sodium chloride solution containing 0.25% riboflavin, I% hydroxyl- propylmethylcellulose, and 0.007% benzalkonium chloride, adjusted to a pH of 7.0, and packaged in 3 mL sterile dropper bottles for topical ophthalmic use. Shelf life is 24 months.

#### 8.3 Supply of Study Drug at Site

The riboflavin solutions will be obtained from: Peschke-MediTrade GmbH Chaesigass 6a 6331 Huenenberg, Switzerland. The study drug is shipped directly to the site. The solution is titled "Peschke-TE (riboflavin 0.25%)":

## 8.4 Storage of Study Drug at Site

The Goodman Eye Center will maintain the experimental study medication in the Laser Room, which is kept locked during non-business hours. It will be stored in a designated cabinet at 68-72 degrees F. The study staff will check the thermometer on Mondays and Wednesdays to ensure that the logs are being completed. The thermometer reads the minimum and maximum temperature for a given day. In the event the temperature is noted to have gone outside of the temperature parameters, the study team will contact the drug provider for guidance immediately. Additionally, the study team will move the product to a back-up refrigerator if needed.

## 8.5 Study Drug Accountability

Study medication (i.e. Riboflavin) will be logged in the Study Drug Dispensing and Inventory Log and will be discarded upon use per clinic and manufacturer guidelines. Unused and expired study drugs will be discarded and disposed per clinic and manufacturer guidelines.

All use of the PXL Platinum 330 Illumination System and Riboflavin 0.25% Ophthalmic Solution will be under the direct supervision of the principal investigator or his designee.

## 8.6 PXL Platinum 330 Illumination System

The PXL Platinum 330 Illumination System is a portable electronic medical device. The device's light emitting diode (LED) is used to deliver a metered dose of UV-A light to a targeted treatment area for illuminating the cornea during corneal collagen cross-linking. Components of the PXL Platinum 330 System include the LED light source, UV light detector, UV detector sensor probe and adapter, wall power supply with DC cord, transportation case, safety goggles (to be worn by user), mechanical stand (C-clamp, cross clamp, rods), and an instruction manual. System specifications are as follows:

Light Source: High Power UV-grade LED; LED Laser class 3R (EN60825-1)

(Mfg. Nichia co. LTD; Tokyo, Japan)

Wavelength: 365 nm (± 10 nm)
Optical Power: Maximum 10 mW
Beam Diameter: 7.5 mm – 11.5 mm
Light Emission: Continuous wave

Intensity Setting: 3.0 mW/cm² (± 0.3 mW/cm²)
Safety Class: Class II Equipment (EN 60601-1)

Medical Device Class: Class IIa according to MDD 93/42/EEC EMI. EMC Class:

Class B (EN 60601-1)

Power Supply: SELV (Safety Extra Low Voltage) 9V; max 1.7A

The *Light Source* houses the UVA irradiation mechanism. The LED is preset by the manufacturer to emit UVA radiation at a wavelength of 365 nm at variable intensities of 3, 9, 18, or 30 mW/cm² (± 0.3 mW/cm). UVA light emission is controlled by an internal microprocessor, which controls the electrical current used to drive the UV-LED. No UV light will be emitted in case of processor or LED failure. The diameter of the Light Source beam aperture is 25 mm and the treatment plane is 50 mm from the beam aperture. An aperture wheel mounted in the UVA irradiation beam path is used to produce a circular area of irradiation at the treatment plane with an approximate diameter of 3 - 12 mm, which is controlled by selecting the corresponding aperture wheel setting on the device. An intensity of 30 mW/cm² and irradiance time of 3 minutes results in a standard surface dose of 5.4 J/cm² surface exposure. With pulsed mode (1 second on, 1 second off), the treatment time doubles. An eye tracker facilitates patient fixation on the light source. The Light Source has an integrated timer that automatically shuts off the light emission after the specified duration

of exposure. A *Power Supply* plugged into a main electrical wall outlet and into the Light Source via the DC cord powers the Light Source. The On/Off switch (On = ready mode) powers the device; the Start/Stop button controls UVA emission; and, status display lights (Red- Internal error, yellow-UV emission, Green-Device is powered, but no UV emission) indicate the status of the PXL Platinum 330 device. A battery operated *UV Light detector*, with a built-in low battery warning, is used to check the UV light irradiation in the treatment plane before patient treatment. The UV Light detector consists of a *Sensor Probe and an indicator*. The *Sensor Probe Adapter* with a Sensor Probe is permanently mounted to the UV-light illumination system to shield the beam aperture and should only be removed for treatment.

#### 9. STUDY VISITS AND PROCEDURES

Prior to any study-related activities, written informed consent, a California Subject's Bill of Rights, and a Health Insurance Portability and Accountability Act (HIPAA) authorization must be signed and dated by the subject or the subject's legal representative. If appropriate, assent must also be obtained prior to conducting any study-related activities.

Demographic, medical, ocular, and medication history of all subjects will be recorded, and the following ophthalmic assessments will be conducted and recorded during the course of the study as further detailed in Appendix A and shown below:

- Demographics
- Contact Lenses History
- Medical History
- Ocular History
- Medication History (Concomitant Medications)
- Uncorrected Visual Acuity (UCVA)
- Manifest Refraction
- Best Corrected Visual Acuity (BCVA)
- Ultrasound Pachymetry
- Pentacam
- Corneal Topography by TMS-4
- Intraocular Pressure (IOP)
- Endothelial Cell Count
- Optical Coherence Tomography K (OCT K)
- Wavefront Aberrometry
- Belin ABCD Progression Display
- Slit Lamp Examination
- Dilated Fundus Exam
- Inclusion/Exclusion Criteria
- Adverse Events

## **Evaluations by Visit**

All subjects will be evaluated at screening (Visit 1) and at randomization/treatment day (Visit 2). Visit 1 and Visit 2 may be combined as one visit. Additional visits will include Day 1 (Visit 3), Day 7/Week 1 (Visit 4), Day 30/Month 1 (Visit 5), Day 90/Month 3 (Visit 6), Day 180/Month 6 (Visit 7), and Day 360/Month 12 (Visit 8).

The study duration is a total of 12 months for all study subjects following the CXL treatment. The duration of the study will also be extended for those subjects who have received retreatment or for subjects who elect to have CXL treatment in an untreated fellow eye.

## 9.1 VISIT 1- Screening Visit (Day -90 to Day 0)

All screening/baseline procedures will be reviewed by the Investigator and/or designee to ensure the subject is appropriate for enrollment. Study candidates who are evaluated preoperatively by referring doctors will sign a study consent form and have the screening procedures repeated preoperatively by the study personnel. Screening data from referring doctors will not be used as the screening data for the study (except the dilated fundus exam if done within the past 12 months) and to document the progression of keratoconus, ectasia, and pellucid marginal degeneration.

Procedures or evaluations that were performed by study personnel during a patient's routine clinic evaluation may be used for screening purposes if the assessments were completed: (1) within 90 days of randomization; (2) in accordance with the protocol requirements; and (3) the screening tests performed are known to be included in the investigator's usual and customary examination procedures. Subjects will sign a consent form before any clinical protocol procedures or tests specific to the study protocol are performed.

After obtaining written informed consent (and assent if appropriate), HIPAA authorization, and Subject Bill of Rights, the following information/assessments will be reviewed and performed as needed, to determine eligibility for study participation:

- Demographics
- History of contact lens wear
- Medical History
- Ocular History (including risk factors for keratoconus)
- Medication History (Concomitant Medications)
- UCVA (distance)
- Manifest Refraction
- BSCVA or best-contacted corrected visual acuity (distance)
- Ultrasound Pachymetry
- Pentacam measurements (including pachymetry, posterior corneal mapping, and keratometry)
- Corneal topography by TMS-4
- IOP (by Goldmann applanation or Tonopen tonometry)
- Endothelial Cell Count (by Cellcheck)
- OCT K

- Wavefront Aberrometry exam by IDesign
- Slit Lamp Examination (of the cornea, anterior chamber, and lens)
- Dilated Fundus Exam
- Inclusion/Exclusion Criteria

For eyes undergoing CXL treatment, if the CXL treatment is performed more than 90 days after any of the screening assessments, those screening assessments will need to be repeated on the day of treatment.

Manifest refractions will be recorded in the source documents in the investigator's usual notation (plus or minus cylinder format). All manifest refractions will be recorded on the case report forms in the study using plus cylinder format.

#### 9.1.1 Contact Lens Discontinuation

Contact Lens wearers should discontinue contact lenses 3 days prior for soft contact lenses or scleral lenses and 2 weeks prior for rigid gas permeable lenses, for their baseline evaluation, treatment, and follow-up visits. Subjects who simply cannot function without wearing their contact lenses have a waiver to the discontinuation regimen.

## 9.1.2 Keratoconus Severity

Eyes that meet the eligibility criteria for progressive keratoconus will be classified according to severity using the grading scheme below adapted from McMahon et al.<sup>34</sup> If the criteria fall into more than one severity category, the severity rating will be based on the keratometry reading. Eyes that are classified as being normal or atypical normal are ineligible for the study and will be recorded as screening failures.

#### Normal

- Regular axial topography pattern (round, oval, symmetric bow tie, etc.)
- Normal slit lamp exam
- o Spectacle corrected acuity 20/20 or better

#### Atypical Normal

- Unusual axial topography explained by slit-lamp exam or history (contact lens warpage, cortical scars not typical of keratoconus, history of refractive surgery)
- Normal or diminished spectacle acuity

## Keratoconus Suspect

- Suspicious axial topography for keratoconus (isolated area of steepening, central steepening > 48 D) but I-S value less than 1.4
- Normal slit lamp exam
- BSCVA 20/20 or better

## Mild Keratoconus

- Axial topography consistent with keratoconus
- Flat keratometry reading < 51.00 D</li>
- Fleischer ring or Vogt striae
- No corneal scarring
- o BSCVA worse than 20/20

#### Moderate Keratoconus

- Axial topography consistent with keratoconus
- Flat keratometry reading between 51.25 D and 56.00 D or astigmatism ≥ 8.00
- Fleischer ring or Vogt striae
- May have corneal scarring up to and including CLEK grade 3.0 (any scarring up to well-defined stromal scarring consistent with keratoconus)
- o BSCVA 20/30 or worse

#### Severe Keratoconus

- Axial topography consistent with keratoconus with marked areas of steepening
- Flat keratometry reading > 56.01 D
- Fleischer ring or Vogt striae
- May have corneal scarring up to and including CLEK grade 4.0 (any scarring up to a dense/opaque stromal scar consistent with keratoconus)
- o BSCVA worse than 20/40

## 9.2 VISIT 2- Procedure Visit (Day 0)

- Medical History
- Ocular History
- Medication History (Concomitant Medications)
- Inclusion/Exclusion Criteria
- Ultrasound Pachymetry
- CXL Treatment and Randomization Procedure
- Ocular Adverse Events
- Schedule subject for Visit 3 in 1-3 days.

## FOLLOW-UP VISITS (POST-PROCEDURE)

## 9.3 VISIT 3- Day 1 Post-Op Visit (1-3 days Post-Op)

- Concomitant Medications
- Ocular Adverse Events
- UCVA
- Slit Lamp Examination
- Schedule subject for Visit 4 in one week (+/- 3 days)

## 9.4 VISIT 4- Day 7/Week 1 Post-Op Visit (+/- 3 days)

- Concomitant Medications
- Ocular Adverse Events
- UCVA
- IOP
- Slit Lamp Examination
- Schedule subject for Visit 5 in one month (+/- 7 days)

## 9.5 VISIT 5- Month 1 Post-Op Visit (+/- 7 days)

- Contact Lenses Information
- Concomitant Medications
- Ocular Adverse Events
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry
- Pentacam
- Corneal topography by TMS-4
- IOP
- Endothelial Cell Count
- OCT K
- Belin ABCD Progression Display
- Slit Lamp Examination
- Schedule subject for Visit 6 in three months (+/- 14 days)

## 9.6 VISIT 6- Month 3 Post-Op Visit (+/- 14 days)

- Contact Lenses History
- Ocular Adverse Events
- Concomitant Medications
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry
- Pentacam
- Corneal topography by TMS-4
- IOP
- Endothelial Cell Count
- Wavefront Aberrometry
- Belin ABCD Progression Display
- Slit Lamp Examination
- Schedule subject for Visit 7 in three months (+/- 30 days)

## 9.7 VISIT 7- Month 6 Post-Op Visit (+/- 30 days)

Contact Lenses History

- Ocular Adverse Events
- Concomitant Medications
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry
- Pentacam
- Corneal topography by TMS-4
- IOP
- Endothelial Cell Count
- OCT K
- Wavefront Aberrometry
- Belin ABCD Progression Display
- Slit Lamp Examination
- Schedule subject for Visit 8 in three months (+/- 30 days)

## 9.8 VISIT 8- Month 12 Post-Op Visit/ End of Study Visit (+/- 30 days)

- Contact Lenses History
- Ocular Adverse Events
- Concomitant Medications
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry
- Pentacam
- Corneal topography by TMS-4
- IOP
- Endothelial Cell Count
- OCT K
- Wavefront Aberrometry
- Belin ABCD Progression Display
- Slit Lamp Examination

Reasonable effort will be made by telephone and mail to contact subjects who miss a scheduled follow-up visit.

## 9.9 Early Withdrawal Visit

- Contact Lenses History
- Ocular Adverse Events
- Concomitant Medications
- UCVA
- Manifest Refraction
- BCVA
- Ultrasound Pachymetry

- Pentacam
- Corneal Topography by TMS-4
- IOP
- Endothelial Cell Count
- OCT K
- Wavefront Aberrometry
- Belin ABCD Progression Display
- Slit Lamp Examination

## 9.10 Early Withdrawal from Study

Subjects will be advised that they are free to withdraw from the study at any time. Subjects experiencing adverse safety events will be followed until the reaction has resolved. Appropriate supportive and/or definitive therapy will be administered as required. The investigator may discontinue a subject if a serious adverse event occurs and it is in the subject's best interest not to continue in the study or if the subject moves and the subject cannot complete the remainder of the follow-up visits. When a subject withdraws early from the study, a final examination will be performed at the time of withdrawal if possible.

#### 10. ADVERSE EVENT REPORTING

## 10.1 Adverse Event Definitions

An adverse event is any untoward and unintended sign, symptom or disease temporrally associated with the use of an investigational drug or other protocol-imposed intervention whether or not considered drug-related.

All treatment-emergent **ocular** adverse events/adverse reactions occurring during the study, and that are not expected and non-serious, should be recorded, regardless of the assumption of causal relationship. Duration (start and stop dates), severity/grade, outcome, treatment, and relation to study treatment will be recorded.

## 10.2 Adverse Event Reporting and Documentation

Eye-related adverse events that are either unexpected and/or serious observed by the Investigator or reported by the subject will be recorded on the study source documents/case report forms. For all adverse events, a description of the event, date first observed, any action taken, and its resolution will be recorded.

## 10.2.1 Expected Non-Serious Ocular Adverse Events

Common and anticipated non-serious adverse events expected to be observed within the first few days and up to four weeks after the procedure and that include the following: pain, photophobia, foreign body sensation, dryness, irritation, and blurred vision, will not be reported to the FDA and/or reported on the subjects case report form.

## 10.3 Classification of Adverse Events by Severity

Severity (intensity) of an adverse event is defined as a qualitative assessment of the level of discomfort of an adverse event as is determined by the Investigator or reported to him/her by the subject. The assessment of intensity is made irrespective of study medication relationship or seriousness of the event and should be evaluated according to the following scale:

**1= Mild:** present, but not distressing, and no disruption of normal daily activity

**<u>2= Moderate:</u>** discomfort sufficient to reduce or affect normal daily activity

3= Severe: incapacitating, with inability to work or perform normal daily activity

A change in severity for a reported AE will require a stop date for the previous severity and a new start and stop date for the new severity. For example, a change in severity might go from mild to moderate or from severe to moderate. In either case, the start and stop dates should be recorded.

## 10.4 Classification of Adverse Event by Relationship

The study medication relationship for each adverse event/adverse reaction should be determined by the Investigator using these explanations:

- **Not Related:** The event is clearly related to other factors such as subject's clinical condition, therapeutic interventions, concomitant disease, therapy administered or accidental trauma of the subject and does not follow a known response pattern to the product.
- Possibly Related: The event follows a reasonable, temporal sequence from
  the time of study medication administration and/or follows a known response
  pattern to the study medication, but could have been produced by other
  factors such as the subject's clinical state, therapeutic interventions or
  concomitant therapy administered to the subject.
- <u>Related:</u> The event follows a reasonable temporal sequence from the time of study medication administration or placement and/or follows a known response pattern to the study medication and cannot be reasonably explained by other factors such as the subject's clinical state, therapeutic interventions or concomitant therapy administered to the subject, and either occurs immediately following study medication administration or there is a positive reaction at the application site.

## 10.5 Serious Adverse Experiences (SAE) Definitions

The sponsor and investigator must comply with the applicable sections of 21CFR312.32 and 21CFR312.64(b) for IND safety reports. In accordance with these regulations, the following definitions apply:

**Associated with the use of the drug**. There is a reasonable possibility that the experience may have been caused by the drug.

**Disability**. A substantial disruption of a person's ability to conduct normal life functions.

**Life-threatening adverse drug experience**. Any adverse drug experience that places the patient or subject, in the view of the investigator, at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction that, had it occurred in a more severe form, might have caused death.

Serious adverse drug experience: Any adverse drug experience occurring at any dose that results in any of the following outcomes: Death, a life-threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Unexpected adverse drug experience: Any adverse drug experience, the specificity or severity of which is not consistent with the current investigator brochure; or, if an investigator brochure is not required or available, the specificity or severity of which is not consistent with the risk information described in the general investigational plan or elsewhere in the current application, as amended. For example, under this definition, hepatic necrosis would be unexpected (by virtue of greater severity) if the investigator brochure only referred to elevated hepatic enzymes or hepatitis. Similarly, cerebral thromboembolism and cerebral vasculitis would be unexpected (by virtue of greater specificity) if the investigator brochure only listed cerebral vascular accidents. "Unexpected," as used in this definition, refers to an adverse drug experience that has not been previously observed (e.g., included in the investigator brochure) rather than from the perspective of such experience not being anticipated from the pharmacological properties of the pharmaceutical product.

## 10.6 Serious Adverse Event Reporting

An investigator shall promptly report to the sponsor any adverse effect that may reasonably be regarded as caused by, or probably caused by, the drug. If the adverse effect is alarming, the investigator shall report the adverse effect immediately.

Any adverse experience associated with the use of the drug that is both serious and unexpected shall be reported by the sponsor to FDA as soon as possible and in no event later than 15 calendar days after the sponsor's initial receipt of the information. Each written notification may be submitted on FDA Form 3500A or in a narrative format and shall bear prominent identification of its contents, i.e., "IND Safety Report." Each written notification to FDA shall be transmitted to the FDA new drug review division in the Center for Drug Evaluation and Research or the product review division in the Center for Biologics Evaluation and Research that has responsibility for review of the IND. If FDA determines that additional data are needed, the agency may require further data to be submitted.

The sponsor shall also notify FDA by telephone or by facsimile transmission of any unexpected fatal or life-threatening experience associated with the use of the drug as soon as possible but in no event later than 7 calendar days after the sponsor's initial receipt of the information. Each telephone call or facsimile transmission to FDA shall be transmitted to the FDA new drug review division in the Center for Drug Evaluation and Research or the product review division in the Center for Biologics Evaluation and Research that has responsibility for review of the IND.

The investigators will promptly report these experiences to the IRB. If the IRB has different or specific reporting deadlines, reports should be made to the IRB in accordance with the IRB's requirements.

## **Serious and Unanticipated Adverse Device Effects**

An unanticipated adverse device effect is defined as "any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, or any other unanticipated serious problem associated with a device that relates to the rights, safety or welfare of subjects." Since CDER has primary jurisdiction for the regulation of this combination product, serious and unanticipated adverse device effects will be reported to FDA and the IRB in accordance with reporting requirements.

## Non-Serious Drug or Device or Anticipated Device Adverse Events

Non-serious and/or unexpected drug or device adverse events and complications should be documented on the case report forms and tabulated for reporting in the annual reports to FDA.

#### 11. PROTOCOL DEVIATIONS

The Investigator will not deviate from the protocol without prior approval from the IRB and the sponsor, unless such deviation is necessary to manage a medical emergency. The investigator will notify the IRB and the sponsor of any protocol deviation to protect the life, ocular health, or physical well-being of a subject in an emergency. Such notice shall be given as soon as possible, but in no event any later than 5 working days after the
emergency occurred. All other revisions and/or amendments to the protocol that affect subject treatment, study outcome, or subject safety will be submitted in writing to the IRB and the sponsor for approval prior to implementation if the changes or deviations to the protocol affect the scientific soundness of the study or the rights, safety, or welfare of human subjects. In this case, the change will not be implemented until IRB approval is obtained. The investigator will maintain a record of all protocol deviations showing the dates of, and the reason for, each protocol deviation.

Changes that affect the scientific soundness of the study or the rights, safety, or welfare of human subjects may also require FDA and IRB approval prior to implementation. The sponsor and investigator will obtain such approvals, if required.

#### 12. DATA ANALYSIS AND STATISTICS

A detailed statistical analysis plan (SAP) will be developed for analysis of all data for this study. The methods by which each of these analyses is performed will be included in the SAP. Required analyses and target endpoints that will be included in this SAP are summarized below.

Tabulation of summary statistics, graphical presentations, and statistical analyses will be performed using RStudio software. All subjects who are enrolled in this study will be included in the safety analysis. All two sided testing and confidence intervals will use a significance level of 5%. The superiority hypotheses will be tested at a significance level of 2.5%.

#### 12.1 Sample Size

The primary efficacy hypothesis for this study, looking at treatment of keratoconus, post-LASIK ectasia, or pellucid marginal degeneration, is to determine whether there is a difference between the two treatment groups in the mean change in best-contact corrected visual acuity (BSCVA) and UCVA compared to the baseline before or after CXL treatment at 3, 6, or 12 months. The null hypothesis is that there is no difference in mean values between the two groups. The data will be analyzed using a two-sample t-test to compare the two treatment groups. The data will be examined using a consistent cohort; therefore patients with missing data (missing post-operative visits) will be excluded from our analysis. This group can also be referred to as the per-protocol (PP) population. All study populations will be defined as intent-to-treat (ITT) populations, however statistical analysis will be performed on the per-protocol population (analysis population), hence excluding the patients with missing post-operative visits.

Since this hypothesis will be tested using a two sample t-test, Figure 12.1-1 presents the sample size (in number of eyes per group) for values obtained from previous studies regarding the difference between the two means, and the standard deviation, with the significance level ( $\alpha$ ) = 0.05 and the power =80%. Previous studies have indicated that the mean baseline UCVA is 20/136 (0.834 logMAR). A difference of 20% between treatment

groups A and B in UCVA is considered to be statistically significant per the investigator. The standard deviation for the differences in UCVA is 0.599 (logMAR)<sup>35</sup>.

It is important to note that the measurements are continuous and therefore the simplest formula for continuous outcomes is implemented in our study<sup>36</sup>. Figure 12.1-1 uses the aforementioned data to calculate sample size for the study.

Figure 12.1-1 Sample Size Calculations for Keratoconus, Ectasia, or PMD Groups

$$nn = \frac{2(1.96 + 0.842)^2(0.599)^2}{(0.667 - 0.834)^2} = 202$$
 eeeeeeeelgggggggggg

Enrolling 202 eyes in each treatment group will enable the detection of a 20% difference in UCVA. We aim to have a minimum of 202 eyes per group to complete the study for both genders.

Since historically there is a 10% discontinuation rate, the sample size is adjusted for a 10% rate of discontinued and lost-to-follow-up eyes:

Adjusted Sample Size (n') = 
$$n/(1-0.10) = n/0.90$$
  
Where n is the initial estimated sample size  
(n') =  $202/0.90$   
(n') =  $224$ 

224 eyes per treatment group (KCN) X 2 genders = 448 eyes

# 12.2 Accountability

Accountability by postoperative visit will be calculated as illustrated in Table 12.2-1 below.

**Table 12.2-1: Accountability by Postoperative Visit** 

| | | 1 Month | 3 Months |
|-------------------------------------|----------|---------|----------|
| Available for Analysis <sup>2</sup> | n/N¹ (%) | | |
| Missed Visit <sup>3</sup> | n/N¹ (%) | | |
| Discontinued <sup>4</sup> | n/N¹ (%) | | |
| Active <sup>5</sup> | n/N¹ (%) | | |
| Lost to follow-up <sup>6</sup> | n/N¹ (%) | | |

| % Accountability = <u>Available for Analysis</u><br>(Enrolled-Discontinued-Active) |
|---|
|---|

#### Where

- <sup>1</sup> Enrolled (N) = total number of subject eyes enrolled in the study.
- <sup>2</sup> Available for analysis = total number of eyes for whom data is available at each postoperative interval.
- <sup>3</sup> Missed visit = total number of eyes that missed the visit, but were otherwise accounted for. Also, includes the eyes that missed the visit but were seen at a later visit.
- <sup>4</sup> Discontinued = total number of eyes that discontinued follow-up prior to completion of the study for any reason (e.g., retreatment, moved away).
- <sup>5</sup> Active (not yet eligible for the interval) = total number of eyes that have not yet reached the visit interval.
- <sup>6</sup> Lost to follow-up = total number of eyes for whom a visit at the prescribed visit or later was not completed and who are not considered to be active or discontinued.

# 12.3 Screening Data

The screening data for all subjects who were screened but did not meet eligibility criteria will not be analyzed or tabulated.

# 12.4 Subject Characteristics

The number of subjects included in the safety and/or effectiveness evaluations, subjects completing the study, and the reasons for any withdrawals will be tabulated by counts and percentages. Continuous demographic data will be summarized using descriptive statistics. Categorical demographic data will be summarized using counts and percentages. Risk factors will be tabulated by eye and summarized using descriptive statistics.

# 12.5 Primary Efficacy Criteria

#### 12.5.1 Visual Acuity

The primary efficacy endpoint of this trial is change in BSCVA or best-contact corrected visual acuity and UCVA compared to the baseline. Study success is defined by the absence of loss of UCVA and BSCVA. All eyes treated (single or both eyes of an individual subject) will be evaluated at each interval postoperatively. Data will be summarized using descriptive statistics. Differences in the mean changes from baseline between the two treatment groups will be tested using a two sample t-test.

As a secondary analysis of this endpoint, a repeated measure analysis of variance will be conducted to assess the profile of the treatments across time at 3, 6, and 12 months.

#### 12.6 Secondary Efficacy Criteria

#### 12.6.1 Keratometry

Secondary efficacy measurements include the corneal curvature, as measured by maximum keratometry ( $K_{max}$ ) and mean keratometry ( $K_{mean}$ ) in the randomized eyes. Study success is defined as the absence of progression of corneal steepening defined as an increase  $K_{max}$  or  $K_{mean}$  of  $\geq 0.5$  diopters from baseline to 12 months in the treated eyes. The change in maximum and mean keratometry ( $K_{max}$  and  $K_{mean}$ ) from baseline will be evaluated at 3 and 12 months. Data will be summarized using descriptive statistics, and the differences in mean changes between Treatment Group A and Treatment Group B will be using a two sample t-test to test the following hypothesis:

$$H_0$$
:CXL - C = 0 versus HA: CXL - C > 0

Where C is the baseline reading ( $K_{max}$  or  $K_{mean}$ ) and CXL is the 3 or 12 month  $K_{max}$  or  $K_{mean}$  reading.

If it assumed the data from both treatment groups are normally distributed, then the test statistic from the ANOVA for testing the above hypothesis is a t-test.

Secondary efficacy measurements will also include: pachymetry, diopters of astigmatism as measured by keratometric cylinder, posterior corneal elevation, manifest refraction, endothelial cell count, and wavefront aberrometry.

#### 12.6.2 Manifest Refraction

The change in the manifest refraction spherical equivalent from baseline will be evaluated at 3 months. Data will be summarized using descriptive statistics. Differences in the mean changes from baseline between the two treatment groups will be tested using a two sample t-test at each time point.

As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 3, 6, and 12 months.

#### 12.6.3 Central Pachymetry

The change in central pachymetry from baseline will be evaluated at 3 months postoperatively. Data will be summarized using descriptive statistics. Differences in the mean changes from baseline between the two treatment groups will be tested using a two sample t-test.

As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 3, 6, and 12 months.

#### 12.6.4 Endothelial Cell Count

The change in endothelial cell density from baseline will be evaluated at 6 months postoperatively. Data will be summarized using descriptive statistics. Differences in the

mean changes from baseline between the two treatment groups will be tested using a two sample t- test at each time point.

As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of treatment across time at 3, 6, and 12 months.

### 12.6.5 Wavefront Aberrometry

The change in wavefront aberrometry, defined as the tabulation of higher order aberrations, will be evaluated at 6 months. Data will be summarized using descriptive statistics. Differences in the mean changes from baseline between the two treatment groups will be tested using a two sample t-test.

As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 3, 6, and 12 months.

# 12.7 Clinical Safety Endpoints

# 12.7.1 Adverse Events and Complications

All subject data, complications, and unexpected and/or serious eye-related adverse events will be tabulated and summarized.

Common expected and non-serious adverse events observed within the first few days and up to four weeks after the procedure that include the following: pain, photophobia, foreign body sensation, dryness, irritation, and blurred vision, will not be reported.

#### 12.7.2 Key Safety Parameters

For each time point, the following key safety parameters will be estimated for the entire cohort.

- 1. Percentage of eyes that had a loss of 2 or more lines in BSCV
- 2. Percentage of eyes that had a BSCVA worse than 20/40
- 3. Percentage of eyes that had a greater than 2D increase in Kmax or Kmean

Safety assessments will also include a tabulation of unexpected and/or serious adverse events, patients symptoms, slit lamp examination of the cornea and lens, and contact lens tolerance for contact lens wearers.

#### 12.8 Dropouts/Lost-to-Follow-Up

Patients may drop out at any time during the study. All treated patients/eyes will be included in the safety analysis.

The primary analysis population for the primary analysis will be based on an Intent-to- Treat population in which missing differences at 3 months for the treatment groups will be

replaced by the smallest maximum difference observed. A per protocol analysis will also be conducted where the missing values are dropped from the analysis.

# 12.9 Interim Analysis

An interim analysis will be performed after all eyes complete the 3-month post-CXL visit. The purpose of this interim analysis is to analyze the safety of the procedure, including all variables tested for at the 3-month interval. All relevant data summaries will be made according to the regulatory process, using appropriate statistical methods. The treatment groups will remain blinded to those performing the post-operative examinations and the interim statistical analysis.

#### 12.10 Sample Size and Randomization

The number of subjects included in the safety and/or effectiveness evaluations, subjects completing the study, and the reasons for any withdrawals will be tabulated by counts and percentages.

#### 13. DATA COLLECTION

#### 13.1 Data Collection Instruments

Adequate records will be maintained for the study including subject medical and surgical records, test reports, work sheets, clinic notes, signed informed consent forms, drug and device use records, adverse experience reports and information regarding subject discontinuation and reasons for discontinuation. All original source documentation will remain at the investigative site. Study data that are stored at the investigator site in any electronic medical record systems, including measurements that are obtained electronically (e.g., pentacam, topography), will be printed and retained in the study files.

All study data will be recorded onto case report forms (electronic or paper) designed for the study. Copies of the case report forms will be retained with the investigator's study files and the original forms will be filed with the sponsor.

#### 14. ADMINISTRATIVE, ETHICAL, REGULATORY CONSIDERATIONS

The study will be conducted in accordance with FDA's Good Clinical Practice regulations.

#### 14.1 Informed Consent

In accordance with the provision of 21 CFR Part 50, each subject will provide written informed consent for participation in this study prior to the use of the investigational device.

The study will be explained to the prospective subject by the Investigator or his designee. The objective of the study will be explained together with potential risks of the procedure, including any possible adverse reactions. The subject will be informed that he/she is free to terminate participation in the study for any reason. A copy of the signed consent form will be given to the subject and the original retained in the Investigator's study chart.

#### 14.2 Institutional Review Board

This protocol and the informed consent form will be approved initially and reviewed annually by an Institutional Review Board (IRB) constituted according to FDA regulations. Progress reports will be submitted at the completion of the study or at least once yearly, whichever comes first, to the IRB. Serious adverse events will be reported to the IRB and the FDA in accordance with applicable FDA regulations for serious adverse events.

#### 14.3 Publications

All manuscripts, abstracts or other modes of presentation arising from the results of the study must be reviewed and approved in writing by the study sponsor in advance of submission.

# 14.4 Investigator Responsibilities

# 14.4.1 Medical and Safety Monitoring

During the CXL treatment procedure, subjects will be observed closely to detect the occurrence of any eye-related adverse events or complications that may have occurred. On the day of treatment and at each follow-up visit, it is suggested that the subjects be asked a non-leading question, such as "How are you seeing?" to determine whether any complications or adverse events might have occurred since the last visit. The presence or absence of adverse events that are unexpected and/or serious, or complications will be documented.

Ophthalmic safety will be evaluated by slit lamp examination of the operated eye, measurements of refraction, and measurement of visual acuity. In the case of an adverse event or complication, these tests may be repeated before the next scheduled visit at the investigator's discretion. Any complications or visual adverse events will be recorded in the medical record/case report form.

Safety monitoring throughout the study will include observations at appropriate times for subjective complaints, complications, eye-related adverse events, clinically significant findings on ophthalmic examination, dilated fundus examination, and slit lamp examination. After treatment, the study subjects will be followed for 12 months total.

# **APPENDIX A: Study Chart Flow**

| Procedure | Screen<br>(Visit #1) | Treatment Visit (Visit #2) | Postoperative Visits | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Day 1<br>(Visit #3)<br>1-3 days<br>Post-Op | Week 1<br>(Visit #4)<br>+/- 3<br>days | Month 1<br>(Visit #5)<br>+/- 7 days | Month 3<br>(Visit #6)<br>+/-14 days | Month 6<br>(Visit #7)<br>+/- 30 days | Month 12<br>(Visit #8)<br>+/- 30 days |
| Informed<br>Consent | X | | | | | | | |
| Demographics | X | | | | | | | |
| History of contact lens wear or corneal infection | X | | | | Х | X | X | Х |
| Medical History | X | X | | | | | | |
| Ocular History | X | X | X | X | Х | X | X | Х |
| Concomitant<br>Meds | X | X | X | X | X | X | X | X |
| UCVA | X | | X | X | X | X | X | Х |
| Manifest<br>Refraction | X | | | | X | X | X | X |
| BCVA | X | | | | Х | X | X | Х |
| Ultrasound<br>Pachymetry | X | X | | | X | X | X | X |
| Pentacam | X | | | | X | X | X | Х |

| Corneal<br>topography by<br>TMS-4 | X | | | | X | X | X | X |
|---|---|---|---|---|---|---|---|---|
| ЮР | X | | | X | X | X | X | Х |
| Endothelial Cell<br>Count | X | | | | X | X | X | X |
| ОСТ К | X | | | | X | | X | X |
| Wavefront<br>Aberrometry | X | | | | | X | X | X |
| Belin ABCD<br>Progression<br>Display | X | | | | X | X | X | X |
| Slit Lamp Exam | X | X | X | X | X | X | X | Х |
| Dilated Fundus<br>Exam | X | | | | | | | X |
| Inclusion<br>Exclusion<br>Criteria | X | X | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X |
| CXL Treatment<br>Randomization<br>and Procedure | | Х | | | | | | |

### **Notes on the Examination Schedule**

- 1.Repeat measurements from the screening exam prior to surgery if needed to provide accurate baseline measurements before CXL treatment.
- 2.Ocular history should include history of contact lens wear, risk factors for keratoconus, and history of refractive surgery. Non-specific questioning should be used at each visit to determine other vision-related complaints, complications, or adverse events
- 3.Distance BCVA should be performed using a Snellen eye chart and recording the total number of letters that are seen
- 4.Distance UCVA should be performed using a Snellen eye chart and recording the total number of letters that are seen
- 5.Intraocular pressure measurement by Goldmann applanation tonometry at a slit lamp or by tonopen.

- 6. The slit lamp exam should include a complete survey of the anterior segment. The cornea should be examined in detail with specific recordings and grading (0 to 4+ scale, 0 = clear) of the following information: overall corneal clarity, any abnormalities such as corneal infiltrates.
- 7.Pentacam measurements are performed using the Pentacam HR (high resolution).
- 8. Endothelial cell count measurements are performed using Konan CellCount.
- 9. Wavefront Aberrometry exam will be performed using IDesign.
- 10.OCT of the cornea will be permed using OptoVue OCT

#### APPENDIX B: CFR 50.25 - Elements of Informed Consent

Basic Elements of Informed Consent: In seeking informed consent, the following information shall be provided to each subject.

- 1. A statement that the study involves research, an explanation of the purpose of the research and the expected duration of the subject's participation, a description of the procedures to be followed, and identification of any procedures which are experimental.
- 2. A description of any reasonably foreseeable risks or discomforts to the subject.
- 3. A description of any benefits to the subject or to others which may reasonably be expected from the research.
- 4. A disclosure of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the subject.
- 5. A statement describing the extent, if any, to which confidentiality of records identifying the subject will be maintained and that notes the possibility that the U.S. Food and Drug Administration may inspect records.
- 6. For research involving more than minimal risk, an explanation as to whether any compensation and an explanation as to whether any medical treatments are available if injury occurs and, if so, what they consist of, or where further information may be obtained.
- 7. An explanation of whom to contact for answers to pertinent questions about the research and research subject's rights, and whom to contact in the event of a research-related injury.
- 8. A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the subject is otherwise entitled, and that the subject may discontinue participation at any time without penalty or loss of benefits to which the subject is otherwise entitled

#### APPENDIX C: World Medical Association Declaration of Helsinki

Ethical Principles for Medical Research Involving Human Subjects Adopted by the 18th WMA General Assembly Helsinki, Finland, June 1964 and amended by the 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 and the 52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### A. INTRODUCTION

- 1. The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.
- 2. It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.
- 3. The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the patient's interest when providing medical care which might have the effect of weakening the physical and mental condition of the patient."
- 4. Medical progress is based on research which ultimately must rest in part on experimentation involving human subjects.
- 5. In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.
- 6. The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic and therapeutic procedures and the understanding of the etiology and pathogenesis of disease. Even the best proven prophylactic, diagnostic, and therapeutic methods must continuously be challenged through research for their effectiveness, efficiency, accessibility and quality.
- 7. In current medical practice and in medical research, most prophylactic, diagnostic and therapeutic procedures involve risks and burdens.
- 8. Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who

- cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.
- 9. Research Investigators should be aware of the ethical, legal and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### B. BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

- 10. It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.
- 11. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.
- 12. Appropriate caution must be exercised in the conduct of research which may affect the environment, and the welfare of animals used for research must be respected.
- 13. The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any serious adverse events. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.
- 14. The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles articulated in this Declaration.
- 15. Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a medically qualified person and never rest on the subject of the research, even though the subject has given consent.

- 16. Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.
- 17. Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.
- 18. Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.
- 19. Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.
- 20. The subjects must be volunteers and informed participants in the research project.
- 21. The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the patient's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.
- 22. In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.
- 23. When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.
- 24. For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law.

These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.

- 25. When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.
- 26. Research on individuals from whom it is not possible to obtain consent, including proxy or advance consent, should be done only if the physical/mental condition that prevents obtaining informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.
- 27. Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 28. The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the patients who are research subjects.
- 29. The benefits, risks, burdens and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic or therapeutic method exists.
- 30. At the conclusion of the study, every patient entered into the study should be assured of access to the best proven prophylactic, diagnostic and therapeutic methods identified by the study.
- 31. The physician should fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study must never interfere with the patient-physician relationship.

32. In the treatment of a patient, where proven prophylactic, diagnostic and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the patient, must be free to use unproven or new prophylactic, diagnostic and therapeutic measures, if in the physician's judgment it offers hope of saving life, reestablishing health or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.

#### **APPENDIX D: References**

- Wollensak, G., Spoerl, E., & Seiler, T. (2003). Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol, 135(5), 620-627.
- Caporossi, A., Baiocchi, S., Mazzotta, C., Traversi, C., & Caporossi, T. (2006). Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italianstudy. J Cataract Reji·act Surg, 32(5), 837-845. doi:J0.10!6/jJcrs.2006.01.091
- 3. Data on File. IROC/University of Dresden. (2006).
- 4. Wollensak, G. (2006). Crosslinking treatment of progressive keratoconus: new hope. Curr Opin Ophthalmol, 17(4), 356-360. doi:10.1097/01.icu.0000233954.86723.25
- Kohlhaas, M., Spoerl, E., Speck, A., Schilde, T., Sandner, D., & Pillunat, L. E. (2005). [A new treatment of keratectasia after LASIK by using collagen with riboflavin/UVA light cross-linking]. Klin Monbl Augenheilkd, 222(5), 430-436. doi:10.1055/s-2005-857950
- 6. Snibson, G. P. I. (2007). A prospective, randomized, clinical trial of corneal collagen cross-linking in progressive keratoconus. Data on File.
- Raiskup, F., Theuring, A., Pillunat, L. E., & Spoerl, E. (2015). Corneal collagen crosslinking with riboflavin and ultraviolet-A light in progressive keratoconus: tenyear results. J Cataract Refract Surg,41(1), 41-46. doi:10.1016/j.jcrs.2014.09.033
- 8. Kumar Kodavoor, S., Arsiwala, A. Z., & Ramamurthy, D. (2014). One-year clinical study on efficacy of corneal cross-linking in Indian children with progressive keratoconus. Cornea, 33(9), 919-922. doi:J0.1097/ico.000000000000197 Labiris
- 9. Vinciguerra, P., Albe, E., Frueh, B. E., Trazza, S., & Epstein, D. (2012). Two-year corneal cross-linking results in patients younger than 18 years with documented progressive keratoconus. Am J Ophthalmol, 154(3),520-526. doi:10.10 i6/j.ajo.2012.03.020
- 10. Vinciguerra, R., Romano, M. R., Camesasca, F. I., Azzolini, C., Trazza, S., Morenghi, E., & Vinciguerra, P. (2013). Corneal cross-linking as a treatment for keratoconus: four- year morphologic and clinical outcomes with respect to patient age. Ophthalmology, 120(5), 908-916. doi:10.1016/j.ophtha.2012.10.023

- 11. Mazzotta, C., Balestrazzi, A., Baiocchi, S., Traversi, C., & Caporossi, A. (2007). Stromal haze after combined riboflavin-UVA corneal collagen cross-linking in keratoconus: in vivo confocal microscopic evaluation. C/in Exp Ophthalmol, 35(6), 580-582. doi:10.111/j.1442-9071.2007.01536.x
- Zamora, K. V., & Males, J. J. (2009). Polymicrobial keratitis after a collagen cross-linking procedure with postoperative use of a contact lens: a case report. Cornea,28(4), 474-476. doi:10.1097/ICO.Ob013e31818d381a
- 13. Vinciguerra, P., Albe, E., Trazza, S., Rosetta, P., Vinciguerra, R., Seiler, T., & Epstein, D. (2009). Refractive, topographic, tomographic, and aberrometric analysis of keratoconic eyes undergoing corneal cross-linking. Ophthalmology, 116(3), 369-378. doi:10.!Ol 6/j.ophtha.2008.09.048
- Caporossi, A., Mazzotta, C., Baiocchi, S., & Caporossi, T. (2010). Long-term results of riboflavin ultraviolet, a corneal collagen cross-linking for keratoconus in Italy: the Siena eye cross study. Am J Ophthalmol,149(4), 585-593. doi:10.10 J6/j.ajo.2009.10.021
- 15. Chatzis, N., & Hafezi, F. (2012). Progression of keratoconus and efficacy of pediatric [corrected] corneal collagen cross-linking in children and adolescents. JRefract Surg, 28(11), 753-758. doi:10.3928/1081597x-20121011-01
- Zotta, P. G., Moschou, K. A., Diakonis, V. F., Kymionis, G. D., Almaliotis, D. D., Karamitsos, A. P., & Karampatakis, V. E. (2012). Corneal collagen cross-linking for progressive keratoconus in pediatric patients: a feasibility study. J Refract Surg, 28(11), 793-799. doi:10.3928/!081597x-2012101!-08
- El Rami, H., Chelala, E., Dirani, A., Fadlallah, A., Fakhoury, H., Cherfan, C., Jarade,
   E. (2015). An Update on the Safety and Efficacy of Corneal Collagen Cross-Linking
   in Pediatric Keratoconus. Biomed Res Int, 2015, 257927. doi:10.1155/2015/257927
- 18. Moramarco, A., Iovieno, A., Sartori, A., & Fontana, L. (2015). Corneal stromal demarcation line after accelerated crosslinking using continuous and pulsed light. J Cataract Reji·act Surg, 41(11), 2546-2551. doi:10.1016/j.jcrs.2015.04.033
- Mazzotta, C., Traversi, C., Caragiuli, S., & Rechichi, M. (2014). Pulsed vs continuous light accelerated corneal collagen crosslinking: in vivo qualitative investigation by confocal microscopy and corneal OCT. Eye (Lond), 28(10), 1179-1183. doi:10.1038/eye.2014.163
- 20. Mazzotta, C., Traversi, C., Paradiso, A. L., Latronico, M. E., & Rechichi, M. (2014). Pulsed Light Accelerated Crosslinking versus Continuous Light Accelerated

- Crosslinking: One-Year Results. J Ophthalmo/, 2014, 604731. doi:10.1155/2014/604731
- 21. Moramarco, A., Iovieno, A., Sartori, A., & Fontana, L. (2015). Corneal stromal demarcation line after accelerated crosslinking using continuous and pulsed light. J Cataract Reji·act Surg, 41(11), 2546-2551. doi:10.1016/j.jcrs.2015.04.033
- 22. Mazzotta, C., Traversi, C., Caragiuli, S., & Rechichi, M. (2014). Pulsed vs continuous light accelerated corneal collagen crosslinking: in vivo qualitative investigation by confocal microscopy and corneal OCT. Eye (Lond), 28(10), 1179-1183. doi:10.1038/eye.2014.163
- Mazzotta, C., Traversi, C., Paradiso, A. L., Latronico, M. E., & Rechichi, M. (2014).
   Pulsed Light Accelerated Crosslinking versus Continuous Light Accelerated
   Crosslinking: One-Year Results. J Ophthalmo/, 2014, 604731.
   doi:10.1155/2014/604731
- 24. www.food.gov.uk/multimedia/pdfs/evm.riboflavin.pdf
- Wollensak, G., Spoerl, E., Reber, F., & Seiler, T. (2004). Keratocyte cytotoxicity of riboflavin/UVA-treatment m vitro. Eye (Lond), 18(7), 718-722. doi:10.1038/sj.eye.6700751
- 26. Wollensak, G., Sporl, E., Reber, F., Pillunat, L., & Funk, R. (2003). Corneal endothelial cytotoxicity of riboflavin/UVA treatment in vitro. Ophthalmic Res, 35(6), 324-328. Doi:74071
- 27. Cho, K. S., Lee, E. H., Choi, J. S., & Joo, C. K. (1999). Reactive oxygen species-induced apoptosis and necrosis in bovine corneal endothelial cells. Invest Ophthalmol Vis Sci, 40(5), 911-919.
- 28. Sporl, E., Schreiber, J., Hellmund, K., Seiler, T., & Knuschke, P. (2000). [Studies on the stabilization of the cornea in rabbits]. Ophthalmologe, 97(3), 203-206.
- 29. Seiler, T. Data on File. IROC.
- 30. Mazzotta, C., Traversi, C., Baiocchi, S., Sergio, P., Caporossi, T., & Caporossi, A. (2006). Conservative treatment of keratoconus by riboflavin-uva-induced cross-linking of corneal collagen: qualitative investigation. Eur J Ophthalmol, 16(4), 530-535.
- 31. Seiler, T., & Hafezi, F. (2006). Corneal cross-linking-induced stromal demarcation line. Cornea, 25(9), 1057-1059. doi:10.1097/01.ico.0000225720.38748.58

- 32. Hafezi, F., Kanellopoulos, J., Wiltfong, R., & Seiler, T. (2007). Corneal collagen crosslinking with riboflavin and ultraviolet A to treat induced keratectasia after laser in situ keratomileusis. J Cataract Refract Surg, 33(12), 2035-2040. doi:10.10 J6/j.jcrs.2007.07.028
- 33. Wittig, C., & Snibson, G. (2007). Aus/rai/ian randomized control trial. Presented at the3rd International Congress of Corneal Cross-Linking, Zurich, Switzerland.
- 34. McMahon, T. T., Szczotka-Flynn, L., Barr, J. T., Anderson, R. J., Slaughter, M. E., Lass, J. H., Group, C. S. (2006). A new method for grading the severity of keratoconus: the Keratoconus Severity Score (KSS). Cornea, 25(7), 794-800. doi:10.1097/01.ico.0000226359.26678.dl
- 35. Noordzij M, Tripep G, Dekker FW, Zoccali C, Tanck MW, Jager KJ. Sample size calculations: basic principles and common pitfalls. Nephrol Dial Transplant (2010) 25: 1388–1393; January 2010
- 36. Stulting RD, Trattler WB, Woolfson JM, Rubinfeld RS. Corneal cross-linking without epithelial removal. Journal of cataract and refractive surgery (2018) 44:1363- 1370; November 2018